CLINICAL TRIAL: NCT04657562
Title: Development and Validation of New LC-MS/MS Method for Determination of Unbound Tacrolimus in Plasma in CYP3A5 Expressors and Non-Expressors
Brief Title: The New LC-MS/MS Method for Determination of Unbound Tacrolimus in Plasma
Acronym: FreeTAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Science Centre, Poland (Other Government)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Karola Warzyszyńska, Medical Doctor, National Science Centre, Poland
Other Study IDs: 2019/33/N/NZ7/01631
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Immunosuppression; Kidney Transplant Rejection; Kidney Transplant; Complications; Liver Transplant Rejection; Liver Transplant; Complications; Metabolism Medication Toxicity; Genetic Predisposition
Keywords: Kidney transplant; liver transplant; CYP3A; unbound tacrolimus; therapeutic drug monitoring
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Blood samples (2 ml and 10 ml test-tubes with EDTA) will be collected to measure
  1. unbound tacrolimus concentration in the human plasma ultrafiltrate
  2. plasma tacrolimus concentration in the human plasma
  3. whole blood tacrolimus through concentration
  4. the DNA will be purified from whole blood and analyzed (RT-PCR).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- De novo renal/liver transplant recipients: The group of 40 consecutive adult (age > 18 years) male and female recipients of deceased kidney or liver transplant from the Regional Qualification Center (Warsaw, Poland).
  Interventions: Drug: Tacrolimus; Diagnostic Test: Unbound tacrolimus measurement; Diagnostic Test: CYP3A4 and CYP3A5 genotyping
- Random renal transplant recipients: The group of 300 random adult (age > 18 years) male and female recipients of deceased kidney attending the local outpatient clinic.
  Interventions: Drug: Tacrolimus; Diagnostic Test: Unbound tacrolimus measurement; Diagnostic Test: CYP3A4 and CYP3A5 genotyping
- Renal transplant recipients experiencing graft rejection: The group of 40 consecutive adult (age > 18 years) male and female recipients of deceased kidney experiencing acute rejection of the renal allograft.
  Interventions: Drug: Tacrolimus; Diagnostic Test: Unbound tacrolimus measurement; Diagnostic Test: CYP3A4 and CYP3A5 genotyping

INTERVENTIONS:
Drug: Tacrolimus — Prevention of rejection in kidney or liver transplant: a standard immunosuppressive therapy according to international protocols.
  Other Names: Prograf; Advagraf
Diagnostic Test: Unbound tacrolimus measurement — Unbound tacrolimus measurement in plasma ultrafiltrate.
Diagnostic Test: CYP3A4 and CYP3A5 genotyping — DNA purification and genotyping

SUMMARY:
Tacrolimus (TAC) is characterized by a narrow therapeutic window, as well as high inter- and intra-individual variability in pharmacokinetics. Both under- and overexposure may lead to severe adverse effects. Therapeutic drug monitoring (TDM) is an essential element of post-transplant patient care. Most transplantation centers use C0 to adjust TAC dosage. Some controversies remain about relationship between C0 and clinical outcome.

It is generally accepted that only protein-unbound drug molecules can cross cellular membranes, which imply that TDM of free tacrolimus fraction may be of paramount importance and improve clinical management of organ recipients.

Whole blood TAC concentrations and dose requirements are strongly associated with CYP3A5 polymorphism. Routine CYP3A5 genotyping on the waiting lists might be useful to guide tacrolimus dosing.

This interdisciplinary project tackles the research problem from three angles - biochemistry, genetics and clinical observation. The primary goal of the study is to evaluate clinical usefulness of different TDM protocols in patients after kidney and liver transplantation.

DETAILED DESCRIPTION:
As there are over 15.000 patients in Poland on continuous tacrolimus (TAC) therapy, the identification and validation of more sensitive and specific biomarkers is of utmost importance. The investigators propose a multiple step assessment of TAC therapeutic drug monitoring (TDM) in kidney and liver recipients. A role of genetic profiling on drug concentration and clinical effects will also be addressed. The project will significantly contribute to understanding tacrolimus pharmacokinetics and body response to drug exposure. Moreover, the proposed project is the first attempt to integrate both different TDM measure methods and patient genetics in a rigorous, prospective study with the assessment of the clinical over- and underexposure TAC effects. It is expected to provide an argument for implementation of even more personalized, predictable immunosuppressive therapy.

The investigators hypothesize that:

1. There is a correlation of free TAC level with drug toxicity on one hand, and graft rejection and underimmunosuppression despite target whole blood concentration on the other.
2. CYP3A5 expressors and non-expressors will present different levels of TAC in both whole blood C0 and free TAC C0 as well as different effectiveness and toxicity profiles.
3. The concentration of free TAC is related to changes in the concentration of blood components, thus it is possible to derive the equation for calculating free TAC concentration as a useful tool for the drug dosage adjustment

Study design

Objectives:

Phase 1) A primary objective of this study is to develop and validate a new method for unbound tacrolimus measurement. - Published: 12 March 2022 (https://doi.org/10.3390/pharmaceutics14030632)

Phase 2) A primary objective is to calculate free fraction of TAC from hematocrit level, albumin concentration and routine whole blood TAC C0 to predict dose adjustment more accurately. The generated equation will be plotted against CYP3A polymorphisms.

Phase 3) A primary objective is to look for a correlation between unbound TAC level in an ultrafiltrate with graft rejection episodes.

Secondary endpoints:

A complex comparison of different methods of determination of TAC concentration in whole blood, plasma and ultrafiltrate is planned.

The benefit of genotyping before administration of TAC for dose prediction will be evaluated.

The studied groups:

1. 40 consecutive kidney or liver transplant recipients on TAC-based immunosuppression.
2. 300 kidney transplant recipients attending the local outpatient clinic.
3. 40 kidney transplant recipients experiencing acute rejection of the renal allograft.

TAC measurements:

Measurements of unbound tacrolimus concentrations in plasma ultrafiltrate and tacrolimus concentrations in plasma and whole blood will be performed using a Nexera LC System with LCMS-8050 MS triple quadrupole with ascomycin and deuterated tacrolimus as internal standards.

Genotyping:

DNA of patients will be purified and analyzed using RT-PCR for CYP3A4 and CYP3A5 polymorphisms Study duration: The study is scheduled for 3 years: 2.5 years for collection of samples, 0.5 year for analysis and publication of the results.

Efficacy variables: Standard monitoring of blood and urine laboratory parameters, whole blood TAC trough level (C0), plasma TAC concentration, free TAC concentration in plasma ultrafiltrate, TAC daily doses.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 yo), recipient of kidney or liver transplant from the Regional Qualification Center, tacrolimus-based immunosuppression

Exclusion Criteria:

* the use of agents significantly influencing TAC metabolism, double organ recipients, HBV, HCV and HIV infection, neurological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. 40 consecutive de novo adult kidney or liver transplant recipients on TAC-based immunosuppression.
  2. 300 adult kidney transplant recipients attending the local outpatient clinic.
  3. 40 adult kidney transplant recipients experiencing acute rejection of the renal allograft.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Development and validation of the new LC-MS/MS measurement method | 1 year
  Development and validation of the extremely sensitive method for unbound tacrolimus determination using the EMA and FDA guidelines
A comparison of different TAC TDM protocols depending on the matrix | 1 year
  1. concentration of unbound tacrolimus in plasma ultrafiltrate
  2. concentration of tacrolimus in plasma
  3. concentration of tacrolimus in whole blood The measures will be obtained with the use of LC-MS/MS method.
Equation to calculate unbound TAC concentration | 1 year
  Development of the equation (using the concentration of free TAC, plasma and whole blood, and blood components) by statistical methods.
A correlation between free TAC and symptoms of underimmunosuppresion | 1 year
  Biopsy proven acute rejection

SECONDARY OUTCOMES:
A correlation between free TAC and nephrotoxicity | 1 year
  Calcineurin inhibitor toxicity confirmed with the biopsy
CYP3A expression | 1 year
  SNP genotyping to address CYP3A genetic variations (CYP3A4 and CYP3A5)
Blood components | 1 year
  Hematocrit, plasma proteins, albumins, LDL, HDL, total cholesterol, triglycerid

CONTACTS AND LOCATIONS:
Overall Officials: Karola Warzyszyńska, MD, Principal Investigator — Department of General and Transplant Surgery, Medical University of Warsaw
Locations (1):
- Department of General and Transplant Surgery, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the study results (about 2023).
Access Criteria: Non-comercial, after request

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Liver transplantation. J Hepatol. 2016 Feb;64(2):433-485. doi: 10.1016/j.jhep.2015.10.006. Epub 2015 Nov 17. No abstract available. PMID 26597456
- [Background] Bittersohl H, Schniedewind B, Christians U, Luppa PB. A simple and highly sensitive on-line column extraction liquid chromatography-tandem mass spectrometry method for the determination of protein-unbound tacrolimus in human plasma samples. J Chromatogr A. 2018 Apr 27;1547:45-52. doi: 10.1016/j.chroma.2018.03.010. Epub 2018 Mar 7. PMID 29544893
- [Background] Brunet M, van Gelder T, Asberg A, Haufroid V, Hesselink DA, Langman L, Lemaitre F, Marquet P, Seger C, Shipkova M, Vinks A, Wallemacq P, Wieland E, Woillard JB, Barten MJ, Budde K, Colom H, Dieterlen MT, Elens L, Johnson-Davis KL, Kunicki PK, MacPhee I, Masuda S, Mathew BS, Millan O, Mizuno T, Moes DAR, Monchaud C, Noceti O, Pawinski T, Picard N, van Schaik R, Sommerer C, Vethe NT, de Winter B, Christians U, Bergan S. Therapeutic Drug Monitoring of Tacrolimus-Personalized Therapy: Second Consensus Report. Ther Drug Monit. 2019 Jun;41(3):261-307. doi: 10.1097/FTD.0000000000000640. PMID 31045868
- [Background] Ekberg H, Tedesco-Silva H, Demirbas A, Vitko S, Nashan B, Gurkan A, Margreiter R, Hugo C, Grinyo JM, Frei U, Vanrenterghem Y, Daloze P, Halloran PF; ELITE-Symphony Study. Reduced exposure to calcineurin inhibitors in renal transplantation. N Engl J Med. 2007 Dec 20;357(25):2562-75. doi: 10.1056/NEJMoa067411. PMID 18094377
- [Background] Pascual J, Berger SP, Witzke O, Tedesco H, Mulgaonkar S, Qazi Y, Chadban S, Oppenheimer F, Sommerer C, Oberbauer R, Watarai Y, Legendre C, Citterio F, Henry M, Srinivas TR, Luo WL, Marti A, Bernhardt P, Vincenti F; TRANSFORM Investigators. Everolimus with Reduced Calcineurin Inhibitor Exposure in Renal Transplantation. J Am Soc Nephrol. 2018 Jul;29(7):1979-1991. doi: 10.1681/ASN.2018010009. Epub 2018 May 11. PMID 29752413
- [Background] Stienstra NA, Sikma MA, van Dapperen AL, de Lange DW, van Maarseveen EM. Development of a Simple and Rapid Method to Measure the Free Fraction of Tacrolimus in Plasma Using Ultrafiltration and LC-MS/MS. Ther Drug Monit. 2016 Dec;38(6):722-727. doi: 10.1097/FTD.0000000000000351. PMID 27805928
- [Background] Bouamar R, Shuker N, Hesselink DA, Weimar W, Ekberg H, Kaplan B, Bernasconi C, van Gelder T. Tacrolimus predose concentrations do not predict the risk of acute rejection after renal transplantation: a pooled analysis from three randomized-controlled clinical trials(dagger). Am J Transplant. 2013 May;13(5):1253-61. doi: 10.1111/ajt.12191. Epub 2013 Mar 8. PMID 23480233
- [Background] Israni AK, Riad SM, Leduc R, Oetting WS, Guan W, Schladt D, Matas AJ, Jacobson PA; DeKAF Genomics Investigators. Tacrolimus trough levels after month 3 as a predictor of acute rejection following kidney transplantation: a lesson learned from DeKAF Genomics. Transpl Int. 2013 Oct;26(10):982-9. doi: 10.1111/tri.12155. Epub 2013 Jul 24. PMID 23879408
- [Background] Kershner RP, Fitzsimmons WE. Relationship of FK506 whole blood concentrations and efficacy and toxicity after liver and kidney transplantation. Transplantation. 1996 Oct 15;62(7):920-6. doi: 10.1097/00007890-199610150-00009. PMID 8878385
- [Background] Zahir H, McCaughan G, Gleeson M, Nand RA, McLachlan AJ. Changes in tacrolimus distribution in blood and plasma protein binding following liver transplantation. Ther Drug Monit. 2004 Oct;26(5):506-15. doi: 10.1097/00007691-200410000-00008. PMID 15385833
- [Background] Zahir H, Nand RA, Brown KF, Tattam BN, McLachlan AJ. Validation of methods to study the distribution and protein binding of tacrolimus in human blood. J Pharmacol Toxicol Methods. 2001 Jul-Aug;46(1):27-35. doi: 10.1016/s1056-8719(02)00158-2. PMID 12164257
- [Background] Hendijani F, Azarpira N, Kaviani M. Effect of CYP3A5*1 expression on tacrolimus required dose for transplant pediatrics: A systematic review and meta-analysis. Pediatr Transplant. 2018 Jun 19:e13248. doi: 10.1111/petr.13248. Online ahead of print. PMID 29920880
- [Background] Rojas L, Neumann I, Herrero MJ, Boso V, Reig J, Poveda JL, Megias J, Bea S, Alino SF. Effect of CYP3A5*3 on kidney transplant recipients treated with tacrolimus: a systematic review and meta-analysis of observational studies. Pharmacogenomics J. 2015 Feb;15(1):38-48. doi: 10.1038/tpj.2014.38. Epub 2014 Sep 9. PMID 25201288
- [Background] Haufroid V, Wallemacq P, VanKerckhove V, Elens L, De Meyer M, Eddour DC, Malaise J, Lison D, Mourad M. CYP3A5 and ABCB1 polymorphisms and tacrolimus pharmacokinetics in renal transplant candidates: guidelines from an experimental study. Am J Transplant. 2006 Nov;6(11):2706-13. doi: 10.1111/j.1600-6143.2006.01518.x. PMID 17049058
- [Background] Venkataramanan R, Swaminathan A, Prasad T, Jain A, Zuckerman S, Warty V, McMichael J, Lever J, Burckart G, Starzl T. Clinical pharmacokinetics of tacrolimus. Clin Pharmacokinet. 1995 Dec;29(6):404-30. doi: 10.2165/00003088-199529060-00003. PMID 8787947
- [Background] Kuypers DR, Claes K, Evenepoel P, Maes B, Vanrenterghem Y. Clinical efficacy and toxicity profile of tacrolimus and mycophenolic acid in relation to combined long-term pharmacokinetics in de novo renal allograft recipients. Clin Pharmacol Ther. 2004 May;75(5):434-47. doi: 10.1016/j.clpt.2003.12.009. PMID 15116056
- [Background] Undre NA, van Hooff J, Christiaans M, Vanrenterghem Y, Donck J, Heeman U, Kohnle M, Zanker B, Land W, Morales JM, Andres A, Schafer A, Stevenson P. Low systemic exposure to tacrolimus correlates with acute rejection. Transplant Proc. 1999 Feb-Mar;31(1-2):296-8. doi: 10.1016/s0041-1345(98)01633-9. No abstract available. PMID 10083114
- [Background] Zong YP, Wang ZJ, Zhou WL, Zhou WM, Ma TL, Huang ZK, Zhao CC, Xu Z, Tan RY, Gu M. Effects of CYP3A5 polymorphisms on tacrolimus pharmacokinetics in pediatric kidney transplantation: a systematic review and meta-analysis of observational studies. World J Pediatr. 2017 Oct;13(5):421-426. doi: 10.1007/s12519-017-0035-4. Epub 2017 May 24. PMID 28540692
- [Background] Nankivell BJ, Alexander SI. Rejection of the kidney allograft. N Engl J Med. 2010 Oct 7;363(15):1451-62. doi: 10.1056/NEJMra0902927. No abstract available. PMID 20925547
- [Background] Randomised trial comparing tacrolimus (FK506) and cyclosporin in prevention of liver allograft rejection. European FK506 Multicentre Liver Study Group. Lancet. 1994 Aug 13;344(8920):423-8. PMID 7520105
- [Background] U.S. Multicenter FK506 Liver Study Group. A comparison of tacrolimus (FK 506) and cyclosporine for immunosuppression in liver transplantation. N Engl J Med. 1994 Oct 27;331(17):1110-5. doi: 10.1056/NEJM199410273311702. PMID 7523946
- [Background] de Mattos AM, Olyaei AJ, Bennett WM. Nephrotoxicity of immunosuppressive drugs: long-term consequences and challenges for the future. Am J Kidney Dis. 2000 Feb;35(2):333-46. doi: 10.1016/s0272-6386(00)70348-9. PMID 10676738
- [Background] Elble R, Comella C, Fahn S, Hallett M, Jankovic J, Juncos JL, Lewitt P, Lyons K, Ondo W, Pahwa R, Sethi K, Stover N, Tarsy D, Testa C, Tintner R, Watts R, Zesiewicz T. Reliability of a new scale for essential tremor. Mov Disord. 2012 Oct;27(12):1567-9. doi: 10.1002/mds.25162. Epub 2012 Oct 2. PMID 23032792